CLINICAL TRIAL: NCT05968105
Title: Evaluation of Lateral Sagittal Infraclavicular Block According to Vena Cava Inferior Collapsibility Index (VCI-CI): An Observational Study
Brief Title: Changes in Vessels After Peripheral Block
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Ergün Mendeş, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Other Study IDs: e.mendes - 3; KAEK/2023.06.260 (Other: Basaksehir Cam and Sakura City Hospital)
Record Dates: First submitted 2023-07-13; First posted 2023-08-01 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Anesthesia, Local; Vena Cava Syndrome (Inferior) (Superior); Fluid Loss; Postoperative Pain
Keywords: Vena Cava Inferior Collapsibility Index; Lateral Sagittal Infraclavicular Block; VCI-CI
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Inferior vena cava diameter <1.5 cm and VCI-CI > 50% according to Vena Cava Inferior Collapsibility Index (VCI-CI)
  Interventions: Procedure: Lateral Sagittal Infraclavicular Block; Diagnostic Test: Inferior vena cava diameter <1.5 cm and Vena Cava Inferior Collapsibility Index (VCI-CI) > 50%
- Group 2: Inferior vena cava diameter >1.5 cm and VCI-CI < 50% according to Vena Cava Inferior Collapsibility Index (VCI-CI)
  Interventions: Procedure: Lateral Sagittal Infraclavicular Block; Procedure: Inferior vena cava diameter >1.5 cm and Vena Cava Inferior Collapsibility Index (VCI-CI) < 50%

INTERVENTIONS:
Procedure: Lateral Sagittal Infraclavicular Block — Patients will be in the supine position and after aseptic conditions are provided, the axillary artery of the patient will be visualized in the craniocaudal plane, in the infraclavicular region and in the lateral sagittal position with the help of an 8-12 mHz linear probe. After the brachial plexus cords around the axillary artery are identified, a local anesthetic mixture will be applied in-plane between the posterior cord and the artery. During the block, patients will routinely be given a mixture of 0.25% bupivacaine + 0.5% lidocaine 0.5 mL/kg.
Procedure: Inferior vena cava diameter >1.5 cm and Vena Cava Inferior Collapsibility Index (VCI-CI) < 50% — While the patients are lying in the supine position, the vena cava will be determined 2 cm before the inferior heart entrance with the help of a 3.5-5 mHz convex probe. M-mode ECHO will be used to determine the fluctuation rate of the VCI between inspiration and expiration. After determining the farthest and closest points in M-mode ECO, their ratios to each other will be calculated.
  Groups: Group 2
Diagnostic Test: Inferior vena cava diameter <1.5 cm and Vena Cava Inferior Collapsibility Index (VCI-CI) > 50% — While the patients are lying in the supine position, the vena cava will be determined 2 cm before the inferior heart entrance with the help of a 3.5-5 mHz convex probe. M-mode ECHO will be used to determine the fluctuation rate of the VCI between inspiration and expiration. After determining the farthest and closest points in M-mode ECO, their ratios to each other will be calculated.
  Groups: Group 1

SUMMARY:
In patients with fluid deficit, vasoconstriction occurs in peripheral tissues and blood circulation is kept in the central area. It causes arterial vasodilation and hemodynamic variability by increasing the blood volume of the extremity due to the sympathectomy occurring after the block. When the investigators classify patients according to VCI-CI, it will be questioned whether there is a difference between patients' block quality and hemodynamic variability.

DETAILED DESCRIPTION:
VCI-CI helps us to have an idea about the amount of fluid in patients according to the vena cava Inferior (VCI) diameter and the diameter between the inspiring and expiration. Low arterial diameter and high inspiratory and expiratory variability indicate that the patient's fluid volume may be lower.

In the measurement of VCI diameter, VCI has visualized in the craniocaudal plane thanks to the transverse ultrasound probe. Changes in VCI diameter are observed depending on the negative pressure in the thoracic area during inspiration and expiration. When the difference between this rate of change is greater than 50%, it indicates that the patient has a fluid deficit. The fact that the VCI diameter is also below 1.5 cm indicates that this amount of fluid requirement is more serious. In this study, the investigators will question whether there is a difference between patients' block quality and hemodynamic variability when they classify patients according to VCI-CI.

ELIGIBILITY:
Inclusion criteria:

* Hand and Wrist elective surgery
* Infraclavicular block will be applied
* American Society of Anesthesiologists (ASA) physical condition I-II
* Patients aged 18-65 years

Exclusion Criteria:

* Contraindication for central or peripheral blocks
* Cognitive dysfunction
* History of chronic opioid use
* severe organ dysfunction
* Allergy to any drug used in the study
* Body mass index (BMI) ≥30
* Infection in the area to be treated
* Refusal to participate in the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Block differences will be observed when patients who undergo routine hand surgery operations under the lateral sagittal infraclavicular block are classified according to the Vena Cava Inferior - Collapsibility Index.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2023-12-03 (Actual); Study Completion 2023-12-03 (Actual)

PRIMARY OUTCOMES:
Doppler flow change from baseline to postoperative period | Perioperative period
  Before the block, with the help of 8-12 mHz linear probe, the axillary artery of the patients will be determined in the lateral sagittal plane and their diameters at the time of systole and diastole will be determined. After the arterial diameters are determined, the probe will be positioned to view the artery in a linear line with 90 degree rotation. After imaging the axillary artery in the long axis, confirming it with 5 sequential flows in B-mode Doppler, PSV (Peak systolic velocity), EDV (End diastolic velocity), mV (mean velocity), RI index and PI index probe angulation at 30-60 degree angle, ultrasound will be measured automatically. After the block, the sensory and motor block times of the patients were determined and these times were recorded.

SECONDARY OUTCOMES:
VAS (Visual Analog Scala) score | Postoperative 24th hour
  The patients were followed up with a VAS score between 0-10 in the postoperative period. A VAS score of 0 was defined as no pain, and 10 as the most severe pain imaginable.
Analgesic consumption | Postoperative 24th hour
  he value in mg of the amount of analgesic consumed in the postoperative period. It was administered with a PCA device that had regular infusions and was able to deliver bolus doses at regular intervals
Postoperative nausea and vomiting | Postoperative 24th hour
  The frequency of nausea and vomiting in the postoperative period was calculated according to the Numeric Rank Score (NRS), which ranged from 0 to 3. Nausea-vomiting status of the patients: 0 points if there is no nausea and vomiting; 1 point if there is nausea, no vomiting; It is scored as 2 points if there is vomiting once and 3 points if there are two or more vomiting attacks.

CONTACTS AND LOCATIONS:
Overall Officials: Ergun Mendes, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Ergun Mendes, Küçükçekmece, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Zhang H, Yuan H, Yu H, Zhang Y, Feng S. Correlation between pleth variability index and ultrasonic inferior vena cava-collapsibility index in parturients with twin pregnancies undergoing cesarean section under spinal anesthesia. Eur J Med Res. 2022 Aug 6;27(1):139. doi: 10.1186/s40001-022-00771-3. PMID 35933431